CLINICAL TRIAL: NCT06586593
Title: ETUDE NEOMEL: TRAITEMENT NEOADJUVANT PAR IMMUNOTHERAPIE DU MELANOME METASTATIQUE OPERABLE EN VIE REELLE (GCC)
Brief Title: Neoadjuvant Immunotherapy of Operable Metastatic Melanoma in Real Life (GCC)
Acronym: NEOMEL
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/758
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Melanoma Metastatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Operable metastatic melanoma: Operable metastatic melanoma

SUMMARY:
This study aims to evaluate efficacy and tolerance of real life neoadjuvant immunotherapy in advanced yet operable melanoma.

The complete histological response will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with operable metastatic melanoma (stage III or IV of American Joint Committee on Cancer [AJCC] Stages CLassification) treated with neoadjuvant immunotherapy (anti-PD1 or anti-PD1 + anti-CTLA-4), even if surgery cancelled due to disease progression or complete response or patient's refusal to be operated.
* Efficacy of the neoadjuvant immunotherapy histologically of radiologically assessed

Exclusion Criteria:

* Uveal melanoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with operable metastatic melanoma (stade III or IV of AJCC) treated with neoadjuvant immunotherapy (anti-PD1 or anti-PD1 + anti-CTLA-4)
Sampling Method: Non-Probability Sample
Enrollment: 77 (Estimated)
Dates: Start 2023-03-24 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Complete histological response | Day 1
  Histological response rate on histological analysis of the resected specimen

SECONDARY OUTCOMES:
Objectival response rate | Day 1
  Objectival response rate on imaging
Event-free survival | Month 12
  An event is defined by progression of the disease or toxicity making surgery impossible, the impossibility of starting adjuvant treatment within 84 days following surgery, recurrence of melanoma after surgery or death.
Disease Free Survival after surgery | Month 12
Overall survival | Month 18
Metastases-free survival | Month 18
Frequency of toxicities | Month 12
  According to Common Terminology Criteria for Adverse Events (CTCAE) v5, grades III and IV
Severity of toxicities | Month 12
  According to CTCAE v5, grades III and IV

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - CHU Angers, Angers
  - CHU de Besançon, Besançon
  - Hôpital Avicenne, Bobigny
  - CH de Boulogne-sur-Mer, Boulogne-sur-Mer
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - Centre de Lutte Contre le Cancer Léon Bérard, Lyon
  - ICO René Gauducheau, Saint-Herblain
  - Institut Universitaire de Cancérologie de Toulouse, Toulouse
  - CH de Valence, Valence

IPD SHARING:
Plan to Share IPD: No